CLINICAL TRIAL: NCT03148873
Title: Evaluation of a Continuous Monitoring Device in Capturing Respiratory Rate Compared to Industry Standard & Gold Standard
Brief Title: RespiraSense Versus Capnography & Manual Counting
Status: Completed | Type: Observational
Sponsor: PMD Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PMD-CS-007
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RespiraSense patient respiratory monitor system — Subjects will have their respiratory rate monitored for two hours using three different methods for capturing it
  Other Names: Capnograph as comparator - Nonin LifeSense Model LS1-9R

SUMMARY:
Your respiratory rate is your number of breaths per minute. The standard way for this to be measured is by a nurse looking at you for one minute and manually counting your breaths over this time. They normally do this once every few hours. At times, it can be useful to have your respiratory rate continuously monitored. A device that can do this is a capnograph. For the patient, this involves wearing a tube in their nose and around their ears while trying to minimise their movement and talking so the measurements can be taken.

This research study is looking at a new respiratory rate monitor and comparing how well it works against the current accepted methods.

Patients who are admitted to the Acute Medical Unit will be invited to participate should they meet all eligibility criteria.

Subjects will be monitored for two hours:

(i) For the first hour subjects will wear a capnograph, RespiraSense and have their respiratory rate manually counted by a research nurse. During this time the subject will be asked to keep talking and moving to a minimum.

(ii) For the second hour subjects will wear RespiraSense and have their respiratory rate manually counted by a research nurse. During this time the subject can talk and move as they wish.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Acute admission to be measured within the first 24 hours of this admission episode
* Are willing to voluntarily sign a statement of informed consent to participate in this investigation

Exclusion Criteria:

* Allergic to medical grade skin adhesive
* Pregnant women during second and third trimester
* Patients who are determined by the medical team to have fragile skin unsuitable for application of the adhesive of the RespiraSense sensor. Patients under the influence of substance abuse (drug or alcohol) that may interfere with their ability to cooperate and comply with the investigation procedures
* Any disorder, including cognitive dysfunction, which would affect the ability to freely give full informed consent
* Patients whose health is deteriorating and unstable
* Patients with predominant palliative care needs
* Patients with a National Early Warning Score (NEWS) of > 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied are patients that have been admitted to the Acute Medical Unit and to be measured within the first 24 hours of this admission episode either on this unit or on whichever ward they have been transferred to.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
RespiraSense versus capnography | 15 minute windows for the first hour of monitoring
  Average respiratory rate

SECONDARY OUTCOMES:
RespiraSense versus manual counting | 15 minute windows for the full two hours of monitoring
  Average respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Christian Subbe, Principal Investigator — BCUHB
Locations (1):
- Ysbyty Gwynedd, Bangor, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No